CLINICAL TRIAL: NCT03637686
Title: Implementing Non-invasive Circulating Tumor DNA Analysis to Optimize the Operative and Postoperative Treatment for Patients With Colorectal Cancer
Brief Title: IMPROVE: Circulating Tumor DNA Analysis to Optimize Treatment for Patients With Colorectal Cancer
Status: Active, not recruiting | Type: Observational
Sponsor: University of Aarhus (Other)
Collaborators: Aarhus University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: IMPROVE
Record Dates: First submitted 2018-07-02; First posted 2018-08-20 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2025-03

CONDITIONS: Colorectal Cancer
Keywords: Colorectal cancer; Circulating tumor DNA
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Tissue Plasma Serum
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The overall objective of these studies are to confirm that ctDNA detected in plasma after intended curative treatment for CRC can be applied in clinical practice as a marker of subclinical residual disease and risk of recurrence.

DETAILED DESCRIPTION:
1. INTRODUCTION Colorectal cancer (CRC) is the third most common cancer worldwide. Approximately two-thirds of patients initially present with potentially curable disease but in spite of curatively intended treatment 30-40% experience relapse of disease. When diagnosed, survival of CRC can basically be improved in two ways, 1) by reducing the risk of recurrence all together, e.g. by improving surgery or by offering adjuvant chemotherapy to the patients with high risk of recurrence, or 2) by early detection of recurrence enabling early intervention which improve patient survival significantly.

   Radical surgery is the most important factor for recurrence and survival of CRC, and free margins of resection are of paramount importance. Initiatives to optimize the quality of surgery, including resection within the correct planes and adherence to the concept of complete mesocolic excision with central ligation of the tumor feeding arteries, are currently being implemented in Denmark. A single Danish center (Hillerød Hospital) which have implemented this technique have reported substantial higher survival rates compared to similar Danish centers using standard surgery.

   Randomized trials have shown that the therapeutic benefit of adjuvant chemotherapy is modest, while the toxicity is substantial. Accordingly, treatment benefit has only been documented for the patients with the highest risk of recurrence (stage III). Nevertheless, also a subset of stage I and stage II patients recur and could potentially benefit from adjuvant therapy. Development of a sensitive approach for assessing if occult residual disease is present after surgery is highly desirable to identify a high-risk sub-group who should be offered adjuvant therapy. Moreover, for stage III disease it is well documented that many patients are overtreated with adjuvant therapy. Surgery alone cures > 40% of such patients and the number needed to treat to prevent a relapse is ~7. Also for these patients, there is need for better and more specific markers of risk of recurrence.

   Solid tumors, including CRC, release DNA fragments into plasma. The plasma of cancer patients contains DNA fragments from both normal and cancer cells. This DNA is referred to as cell free DNA (cfDNA), while the specific fraction that originates from tumor cells is called circulating tumor DNA (ctDNA). The investigators have recently presented results that, in line with others, indicate that patients with ctDNA detected post-surgery are at extremely high risk of a later radiologic recurrence (HR=37.66; 95% CI, 4.23 to 335.49; P<0.0001). This risk is greater than that in patients with stage III colorectal cancer who are routinely treated with adjuvant therapy. These findings show that post-operative ctDNA analysis has potential to become a highly valuable tool for assessment of the quality of the primary surgery and for guiding the use of adjuvant therapy.

   In agreement with others, the investigators have shown that ctDNA changes detected through longitudinal analysis correlates closely with changes in tumor volume as assessed by CT-imaging. Thus, ctDNA analysis has potential as a tool for assessing the impact of intervention (e.g. chemotherapy, surgery, radio frequency ablation (RFA), and stereotactic body therapy (SRBT)). The investigators have shown that serial ctDNA analysis enable detection of incipient clinical disease recurrence on average 10 months before by the conventional modalities (primarily CT-scan. Accordingly, ctDNA analysis has the potential to provide a critical window of opportunity for intervention at an early time-point where curative modalities are still an option.
2. INVESTIGATIONAL PLAN 2.1 Overall study design The IMPROVE - OBSERVATIONAL STUDIES are based on a comprehensive series of blood sampling and ctDNA analysis performed in CRC patients before and after surgery, during and after adjuvant chemotherapy, and during surveillance. Patients are followed 5 years from date of surgery.

The IMPROVE OBSERVATIONAL STUDIES logistically consist of two parts:

IMPROVE OBSERVATIONAL STUDY PART I - SURGERY This part comprises blood sampling and ctDNA analysis pre-operative and immediately after surgery (post-OP day 14) and sampling of tissue from the resected specimen.

IMPROVE OBSERVATIONAL STUDY PART II - SURVEILLANCE This part comprises longitudinal blood sampling over a 5 year surveillance period.

IMPROVE INTERVENTIONAL STUDY - IMPROVE IT A subset of patients included in IMPROVE PART I - SURGERY are candidates for inclusion in the IMPROVE INTERVENTIONAL STUDY - IMPROVE IT. The IMPROVE IT study is described in detail in a separate protocol.

2.2 Sample size We will include at least 1800 patients treated with curative intend for stage I-III disease. We have recently reported a study showing that ctDNA was detectable in plasma (drawn shortly after surgery) from 57% of relapsing stage II and III patients and in 0% of the non-relapse patients. In the present study, we expect a higher sensitivity as we will be analyzing ~8 times larger blood volumes than previously. We expect the following stage distribution: stage I, 28%; stage II, 37%; stage III, 35%9; and estimated ~223 relapse events (expected relapse rates: stage I, 7%; stage II, 12%; stage III, 17%). When combining our previous results with the size of the suggested cohort and with the expected distribution and relapse events, this translates into a power of >99.9% at a precision level of 1% (two-tailed) for confirming prognostic significance of ctDNA at the end of the study.

2.3 Collection of biological samples (Blood and tissue) 2.3.1 Time points for sample collection - IMPROVE PART I -SURGERY For all patients included in part I (Surgery) blood samples will be drawn prior to and after surgery. Whenever possible fresh tumor and adjacent normal mucosa biopsies will be collected from the surgical resected specimen, otherwise formalin-fixed paraffin-embedded tissues will be obtained from the archives.

2.3.2 Time points for sample collection - IMPROVE PART II - SURVEILLANCE For all patients included in part II (surveillance) blood samples will be drawn longitudinally during the post-surgical follow-up period: three times in year 1, three times in year 2, twice in year 3, and once a year in years 4 and 5.

2.3.3 Time point for identification of candidates for IMPROVE IT. The candidates are patients with stage I or II disease and WITHOUT risk factors qualifying for adjuvant chemotherapy, and who's day 14 blood sample is ctDNA positive. Patients that consented to receive the day 14 blood sample result are approached and invited to participate in IMPROVE-IT. Before inclusion the patients are offered a PET-CT scan, to ensure that no metastases have been overlooked.

If the day 14 sample is ctDNA negative the patients are informed that their relapse risk is low and that they will receive surveillance according to DCCG guidelines.

Patients with indications for adjuvant chemotherapy are informed that they will NOT receive information about the analysis results of their day 14 blood sample, since this will not change their planned treatment course. The patients are asked to consent to longitudinal blood sampling and ctDNA analysis (inclusion in IMPROVE PART II - SURVEILLANCE), no matter whether they will receive adjuvant chemotherapy or not.

2.4 Molecular analysis 2.4.1 Detection and quantification of circulating tumor DNA Detection and quantification of ctDNA will be performed using our recently developed ultra-sensitive targeted duplex sequencing approach. Using this approach, we will sequence more than 5,000 unique DNA molecules from each plasma sample. Thereby, detection of somatic mutations with allele frequencies down to ~0.1% is possible. Further, our improved method includes multiple steps aimed at reducing the error rate, including the use of unique strand-specific molecular barcodes (UMIs) and redundant sequencing of each cfDNA fragment. Thereby we can distinguish polymerase induced errors from true mutations.

The sequencing approach targets <100.000 of the 3 billion bases in the human genome. The panel comprise the most common and important CRC driver mutations identified in the IntOGEN and TCGA databases. Multiple redundant capture probes are used for each gene to improve coverage and provide higher specificity. Targeting these regions is sufficient to ensure that at least one somatic mutation will be identified in each CRC case and should therefore enable assessment of the ctDNA level in all included patients. The gene regions included in the panel are: TP53 exon 5-8 (1792 bases), KRAS codons 12, 13, 61, 117, and 146 (738 bases), SMAD2 selected frequently mutated regions (463 bases), SMAD4 selected frequently mutated regions (513 bases), FAM123B selected frequently mutated regions (669 bases), SOX9 selected frequently mutated regions (693 bases), APC selected frequently mutated regions (5477 bases), TCF7L2 selected frequently mutated regions (920 bases), NRAS codons 12, 13, and 61 (405 bases), BRAF codon 600 and others nearby (200 bases), FBXW7 selected frequently mutated regions (868 bases), PIK3CA 8 hotspot mutations (905 bases).

2.5 Collection of clinical Information A central part of the project involves comparison and correlation of the ctDNA assessments (gathered from the blood samples) with the clinical information on treatment and outcome. Clinical information regarding the treatment and outcome of the treatment will be collected from hospital records and health registries.

2.6 Definitions of predictor variables, co-variates and end-points 2.6.1 Primary endpoint

* Disease free survival at 3 years (3y-DFS) 2.6.2 Secondary endpoints
* Local and/or distant recurrence (pathological, radiological or clinical)
* Time to recurrence (TTR)
* Disease free survival at 1 year (1y-DFS))
* Overall survival at year 5 (5y-OS)
* Molecular residual disease
* Time to molecular recurrence (TTMR) 2.6.3 Safety Endpoint
* Frequency and severity of adverse events (AE) in relation to the per protocol blood draws.

2.6.4 Definition of endpoints

* DFS is defined as the time from surgery to the first occurrence of any of the following events; loco-regional recurrence, distant metastases, or death from any cause.
* Time to recurrence is calculated from date of surgery until loco-regional recurrence or distant metastases, or death from colorectal cancer.
* Overall survival is defined as the time from surgery to death from any cause.
* Molecular residual disease is defined as detection of circulating tumor DNA (ctDNA) in a blood sample drawn shortly after the end of a curatively intended treatment (between day 1 and day 30 post-surgery, or between day 1 and day 30 after end of adjuvant therapy).
* Time to molecular recurrence is calculated from first time of no detectable ctDNA until detectable ctDNA.

2.7 Statistical analysis 2.7.1 Analysis of DFS, OS, TTR Kaplan-Meier estimates will be used for the estimation of median times to recurrence (clinical and molecular), disease or death and their confidence intervals, stratified according to UICC stage and/or post-OP ctDNA status. Endpoints will be assessed using the log-rank test or a Cox regression model, with time to event (clinical or molecular recurrence or death) as response variable and ctDNA post-surgery or adjuvant therapy as factor.

ELIGIBILITY:
Part I: Surgery

Inclusion Criteria:

* Colon or rectal cancer, clinical tumor stage I-III
* Patient able to understand and sign written informed consent
* Scheduled for curative intended resectional surgery

Exclusion Criteria:

* Hereditary colorectal cancer linked to familial colonic polyposis or Lynch syndrome
* Inflammatory bowel disease (Crohn's disease or ulcerative colitis)
* Verified distant metastases
* Malignant colorectal polyps diagnosed after polypectomy
* Patients who are unlikely to comply with the protocol (e.g. uncooperative attitude, inability to return for subsequent visits) and/or otherwise considered by the Investigator to be unlikely to complete the study

Part II: Surveillance:

Inclusion criteria:

One of the following:

* TNM stage III CRC,
* or TNM stage II CRC and risk factors qualifying for adjuvant chemotherapy,
* or TNM stage I or stage II CRC without risk factors, but ctDNA positive in the post-operative day14 plasma sample. Inclusion requires that the patient declined participation in the IMPROVE IT trial.

Exclusion criteria:

* Synchronous colorectal and non-colorectal cancer diagnosed per-operative (except skin cancer other than melanoma)
* Other cancers (excluding colorectal cancer or skin cancer other than melanoma) within 3 years from screening

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients with stage I-III colon or rectal cancer, scheduled for curative intended resectional surgery.
Sampling Method: Probability Sample
Enrollment: 3182 (Actual)
Dates: Start 2018-06-14 (Actual); Primary Completion 2028-07-01 (Estimated); Study Completion 2035-07-01 (Estimated)

PRIMARY OUTCOMES:
Patients with high risk of recurrence can be identified with ctDNA profiling performed immediately after treatment for CRC. | 3 years
  3-year disease-free survival (3y-DFS)

SECONDARY OUTCOMES:
Association between ctDNA and the quality of primary surgery - the plane of the surgery | 3 years
  Association between presence of ctDNA measured by sequencing cfDNA and the plane of the surgery in the pathological specimen (muscular, intrameso-colic/rectal, meso-colic/rectal)
Association between ctDNA and the quality of primary surgery - the level of resection of the tumor feeding arteries | 1 years
  Association between presence of ctDNA measured by sequencing cfDNA and the length of the feeding artery in the resection specimen and the length of the artery residue in the patient measured on the first follow-up CT scan (at 12 month post-OP), respectively.
ctDNA profiling for evaluating quality improvement of surgery - before and after implementation of of a training program | 3 years
  ctDNA is measured by sequencing cfDNA. The rate of detection of ctDNA post-operatively is compared between resections performed before and after implementation of the training program at five Danish surgical centers.
ctDNA profiling for evaluating quality improvement of surgery - between centers with and without implementation of the training program | 3 years
  ctDNA is measured by sequencing cfDNA. The rate of detection of ctDNA post-operatively is compared between resections performed at centers with and without implementation of the training program.
Association between ctDNA and the effect of adjuvant chemotherapy | 3 years
  ctDNA measured by sequencing cfDNA. ctDNA measurements are performed before and after adjuvant chemotherapy. Changes in ctDNA level will be correlated to oncological outcome by measuring time to clinical recurrence, disease-free survival and overall survival.
Can ctDNA detect recurrence earlier than standard-of-care? | 7 years
  The difference between time to molecular recurrence (ctDNA detection) is compared to the time to clinical recurrence measured on CT scans..

CONTACTS AND LOCATIONS:
Overall Officials: Claus L Andersen, PhD, Principal Investigator — University of Aarhus; Søren Laurberg, MD, PhD, Principal Investigator — Aarhus University Hospital; Karen-Lise G Spindler, MD, PhD, Principal Investigator — Aarhus University Hospital
Locations (10):
- Denmark (10):
  - Aalborg University Hospital, Aalborg, North Denmark
  - Odense University Hospital, Odense, The Region of Southern Denmark
  - Aarhus University Hospital, Aarhus
  - Bispebjerg Hospital, Copenhagen
  - Herlev Hospital, Herlev
  - Regional Hospital West Jutland, Herning
  - Regional Hospital Horsens, Horsens
  - Zealand University Hospital, Køge
  - Regional Hospital Randers, Randers
  - Regional Hospital Viborg, Viborg

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Scholer LV, Reinert T, Orntoft MW, Kassentoft CG, Arnadottir SS, Vang S, Nordentoft I, Knudsen M, Lamy P, Andreasen D, Mortensen FV, Knudsen AR, Stribolt K, Sivesgaard K, Mouritzen P, Nielsen HJ, Laurberg S, Orntoft TF, Andersen CL. Clinical Implications of Monitoring Circulating Tumor DNA in Patients with Colorectal Cancer. Clin Cancer Res. 2017 Sep 15;23(18):5437-5445. doi: 10.1158/1078-0432.CCR-17-0510. Epub 2017 Jun 9. PMID 28600478
- [Background] Reinert T, Scholer LV, Thomsen R, Tobiasen H, Vang S, Nordentoft I, Lamy P, Kannerup AS, Mortensen FV, Stribolt K, Hamilton-Dutoit S, Nielsen HJ, Laurberg S, Pallisgaard N, Pedersen JS, Orntoft TF, Andersen CL. Analysis of circulating tumour DNA to monitor disease burden following colorectal cancer surgery. Gut. 2016 Apr;65(4):625-34. doi: 10.1136/gutjnl-2014-308859. Epub 2015 Feb 4. PMID 25654990
- [Background] Phallen J, Sausen M, Adleff V, Leal A, Hruban C, White J, Anagnostou V, Fiksel J, Cristiano S, Papp E, Speir S, Reinert T, Orntoft MW, Woodward BD, Murphy D, Parpart-Li S, Riley D, Nesselbush M, Sengamalay N, Georgiadis A, Li QK, Madsen MR, Mortensen FV, Huiskens J, Punt C, van Grieken N, Fijneman R, Meijer G, Husain H, Scharpf RB, Diaz LA Jr, Jones S, Angiuoli S, Orntoft T, Nielsen HJ, Andersen CL, Velculescu VE. Direct detection of early-stage cancers using circulating tumor DNA. Sci Transl Med. 2017 Aug 16;9(403):eaan2415. doi: 10.1126/scitranslmed.aan2415. PMID 28814544